CLINICAL TRIAL: NCT02410447
Title: Defocused Shock Wave Therapy for Chronic Soft Tissue Wounds of the Lower Limbs. A Pilot Study
Brief Title: Defocused Shock Wave Therapy for Chronic Wounds
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Mario Vetrano, MD, MD, University of Roma La Sapienza
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2
Record Dates: First submitted 2015-03-27; First posted 2015-04-07 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Wounds
Keywords: Shock waves
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Group (Experimental): Defocused shock waves were provided by an electromagnetic generator (DUOLITH® SD1 - Storz Medical AG, Tägerwilen, Switzerland).
  The protocol consisted of a series of 3 sessions in 2 weeks, 2 treatments a week. For each patient, a different number of impulses per session was delivered, depending on wound size (300 impulses + 100 impulses per cm2 wound-surface), at an energy flux density of 0.15 mJ/mm2 and a frequency of 5 pulses/s.
  Interventions: Device: Defocused shock wave therapy (DUOLITH® SD1)

INTERVENTIONS:
Device: Defocused shock wave therapy (DUOLITH® SD1)

SUMMARY:
Chronic soft tissue wounds of the lower limbs are painful and debilitating condition that significantly reduce the quality of life of the patient. They often do not respond to conservative treatments or advanced wound managements. Focused and defocused extracorporeal shock wave therapy can be a viable alternative therapeutic strategy.

The purpose of the study was to examine the effects of defocused extracorporeal shock wave treatment on chronic soft tissue wounds of the lower limbs, in terms of the rate of wound healing and pain control.

ELIGIBILITY:
Inclusion Criteria:

* chronic post-traumatic, venous, arterial, diabetic, or mixed wound of the lower limb
* wound persisting for longer than three months
* a wound surface bigger than 0,5 cm2
* a wound diameter between 0.5 and 5 cm
* unresponsiveness to conservative treatments and advanced wound managements in the 3 months prior to enrollment
* no changes in wound managements during the study.

Exclusion Criteria:

* an ankle brachial index (ABPI)<0.7 and TcPO2<40 mmHg
* arrhythmias, presence of pacemaker, or coagulation disorders
* use of anticoagulant drugs
* neoplasia
* pregnancy
* soft tissue wound infections and/or osteomyelitis
* patients with full-thickness loss of soft tissue and extension into muscle, bone, tendon, or joint capsule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-05; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Changes from baseline of the wound surface | 15 days, 1 month and 3 months after treatment
  Computerized digital photo documentation was used to define the size of the wound with a specific software

SECONDARY OUTCOMES:
Changes from baseline of the wound characteristic | 15 days, 1 month and 3 months after treatment
  Wounds characteristics were assessed by the Bates-Jensen Wound Assessment Tool
Improvement in subjective wound-related pain intensity | 15 days, 1 month and 3 months after treatment
  Subjective wound-related pain was evaluated using the Visual Analogue Score

CONTACTS AND LOCATIONS:
Locations (1):
- Sant'Andrea Hospital, Rome, Italy, Italy

REFERENCES:
- [Background] Schaden W, Thiele R, Kolpl C, Pusch M, Nissan A, Attinger CE, Maniscalco-Theberge ME, Peoples GE, Elster EA, Stojadinovic A. Shock wave therapy for acute and chronic soft tissue wounds: a feasibility study. J Surg Res. 2007 Nov;143(1):1-12. doi: 10.1016/j.jss.2007.01.009. Epub 2007 Sep 27. PMID 17904157
- [Background] Saggini R, Figus A, Troccola A, Cocco V, Saggini A, Scuderi N. Extracorporeal shock wave therapy for management of chronic ulcers in the lower extremities. Ultrasound Med Biol. 2008 Aug;34(8):1261-71. doi: 10.1016/j.ultrasmedbio.2008.01.010. Epub 2008 Apr 18. PMID 18394777
- [Background] Moretti B, Notarnicola A, Maggio G, Moretti L, Pascone M, Tafuri S, Patella V. The management of neuropathic ulcers of the foot in diabetes by shock wave therapy. BMC Musculoskelet Disord. 2009 May 27;10:54. doi: 10.1186/1471-2474-10-54. PMID 19473538
- [Background] Arno A, Garcia O, Hernan I, Sancho J, Acosta A, Barret JP. Extracorporeal shock waves, a new non-surgical method to treat severe burns. Burns. 2010 Sep;36(6):844-9. doi: 10.1016/j.burns.2009.11.012. Epub 2010 Jan 13. PMID 20071091
- [Background] Mittermayr R, Antonic V, Hartinger J, Kaufmann H, Redl H, Teot L, Stojadinovic A, Schaden W. Extracorporeal shock wave therapy (ESWT) for wound healing: technology, mechanisms, and clinical efficacy. Wound Repair Regen. 2012 Jul-Aug;20(4):456-65. doi: 10.1111/j.1524-475X.2012.00796.x. Epub 2012 May 29. PMID 22642362
- [Background] Haupt G, Chvapil M. Effect of shock waves on the healing of partial-thickness wounds in piglets. J Surg Res. 1990 Jul;49(1):45-8. doi: 10.1016/0022-4804(90)90109-f. PMID 2359293
- [Background] Kuo YR, Wang CT, Wang FS, Yang KD, Chiang YC, Wang CJ. Extracorporeal shock wave treatment modulates skin fibroblast recruitment and leukocyte infiltration for enhancing extended skin-flap survival. Wound Repair Regen. 2009 Jan-Feb;17(1):80-7. doi: 10.1111/j.1524-475X.2008.00444.x. PMID 19152654
- [Background] Wang CJ, Wu RW, Yang YJ. Treatment of diabetic foot ulcers: a comparative study of extracorporeal shockwave therapy and hyperbaric oxygen therapy. Diabetes Res Clin Pract. 2011 May;92(2):187-93. doi: 10.1016/j.diabres.2011.01.019. Epub 2011 Apr 6. PMID 21310502
- [Background] Mariotto S, Cavalieri E, Amelio E, Ciampa AR, de Prati AC, Marlinghaus E, Russo S, Suzuki H. Extracorporeal shock waves: from lithotripsy to anti-inflammatory action by NO production. Nitric Oxide. 2005 Mar;12(2):89-96. doi: 10.1016/j.niox.2004.12.005. PMID 15740982
- [Background] Ohtori S, Inoue G, Mannoji C, Saisu T, Takahashi K, Mitsuhashi S, Wada Y, Takahashi K, Yamagata M, Moriya H. Shock wave application to rat skin induces degeneration and reinnervation of sensory nerve fibres. Neurosci Lett. 2001 Nov 23;315(1-2):57-60. doi: 10.1016/s0304-3940(01)02320-5. PMID 11711214
- [Background] Kuo YR, Wang CT, Wang FS, Chiang YC, Wang CJ. Extracorporeal shock-wave therapy enhanced wound healing via increasing topical blood perfusion and tissue regeneration in a rat model of STZ-induced diabetes. Wound Repair Regen. 2009 Jul-Aug;17(4):522-30. doi: 10.1111/j.1524-475X.2009.00504.x. PMID 19614917
- [Background] Hayashi D, Kawakami K, Ito K, Ishii K, Tanno H, Imai Y, Kanno E, Maruyama R, Shimokawa H, Tachi M. Low-energy extracorporeal shock wave therapy enhances skin wound healing in diabetic mice: a critical role of endothelial nitric oxide synthase. Wound Repair Regen. 2012 Nov-Dec;20(6):887-95. doi: 10.1111/j.1524-475X.2012.00851.x. Epub 2012 Oct 30. PMID 23110611
- [Background] Larking AM, Duport S, Clinton M, Hardy M, Andrews K. Randomized control of extracorporeal shock wave therapy versus placebo for chronic decubitus ulceration. Clin Rehabil. 2010 Mar;24(3):222-9. doi: 10.1177/0269215509346083. Epub 2010 Feb 15. PMID 20156981
- [Background] Stieger M, Schmid JP, Bajrami S, Hunziker T. [Extracorporeal shock wave therapy as a treatment of a non-healing chronic leg ulcer]. Hautarzt. 2013 Jun;64(6):443-6. doi: 10.1007/s00105-012-2527-4. German. PMID 23322179
- [Background] Omar MT, Alghadir A, Al-Wahhabi KK, Al-Askar AB. Efficacy of shock wave therapy on chronic diabetic foot ulcer: a single-blinded randomized controlled clinical trial. Diabetes Res Clin Pract. 2014 Dec;106(3):548-54. doi: 10.1016/j.diabres.2014.09.024. Epub 2014 Oct 5. PMID 25451894
- [Background] Wolff KS, Wibmer A, Pusch M, Prusa AM, Pretterklieber M, Teufelsbauer H, Schaden W. The influence of comorbidities and etiologies on the success of extracorporeal shock wave therapy for chronic soft tissue wounds: midterm results. Ultrasound Med Biol. 2011 Jul;37(7):1111-9. doi: 10.1016/j.ultrasmedbio.2011.04.007. Epub 2011 Jun 2. PMID 21640475
- [Background] Wang CJ, Kuo YR, Wu RW, Liu RT, Hsu CS, Wang FS, Yang KD. Extracorporeal shockwave treatment for chronic diabetic foot ulcers. J Surg Res. 2009 Mar;152(1):96-103. doi: 10.1016/j.jss.2008.01.026. Epub 2008 Mar 7. PMID 18619622